CLINICAL TRIAL: NCT03260491
Title: A Multicenter, Open-Label Phase 1 Study of U3-1402 in Subjects With Metastatic or Unresectable Non-small Cell Lung Cancer
Brief Title: U3-1402 in Metastatic or Unresectable Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-U102; 2024-511205-33-00 (EU CTIS Number); 194868 (Other: JapicCTI)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Oncology; Advanced Non-small Cell Lung Cancer; Metastatic; Unresectable; Epidermal growth factor receptor; EGFR; KRAS-G12C; Unresectable Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Dose Escalation: Cohort 1, 3.2 mg/kg (Experimental): Participants in the Dose Escalation Cohort 1 will receive HER3-DXd intravenously (IV) once every three weeks at 3.2 mg/kg.
  Interventions: Drug: HER3-DXd (FL-DP)
- Dose Escalation: Cohort 2, 4.8 mg/kg (Experimental): Participants in Dose Escalation Cohort 2 will receive HER3-DXd intravenously (IV) once every three weeks at 4.8 mg/kg.
  Interventions: Drug: HER3-DXd (FL-DP)
- Dose Escalation: Cohort 3, 5.6 mg/kg (Experimental): Participants in Dose Escalation Cohort 3 will receive HER3-DXd intravenously (IV) once every three weeks at 5.6 mg/kg.
  Interventions: Drug: HER3-DXd (FL-DP)
- Dose Escalation: Cohort 4, 6.4 mg/kg (Experimental): Participants in Dose Escalation Cohort 3 will receive HER3-DXd intravenously (IV) once every three weeks at 6.4 mg/kg.
  Interventions: Drug: HER3-DXd (FL-DP)
- Dose Expansion: Cohort 1, EGFR mutant (Experimental): Participants with adenocarcinoma NSCLC with EGFR mutations in the Dose Expansion Cohort 1 will receive HER3-DXd IV once every three weeks at the established recommended dose for expansion (RDE).
  Interventions: Drug: HER3-DXd (CTM-1 Lyo-DP)
- Dose Expansion: Cohort 2, EGFR wild-type (Experimental): Participants with squamous or non-squamous NSCLC without EGFR-activating mutations in the Dose Expansion Cohort 2 will receive HER3-DXd IV once every three weeks at the established recommended dose for expansion (RDE).
  Interventions: Drug: HER3-DXd (CTM-1 Lyo-DP)
- Dose Expansion: Cohort 3a, EGFR mutant (Experimental): Randomized participants with NSCLC and EGFR mutations in the Dose Expansion Cohort 3a will receive HER3-DXd IV once every three weeks at the established recommended dose for expansion (RDE) or, if applicable, adjusted RDE (aRDE).
  Interventions: Drug: HER3-DXd (CTM-1 Lyo-DP)
- Dose Expansion: Cohort 3b, EGFR mutant (Experimental): Randomized participants with NSCLC and EGFR mutations in the Dose Expansion Cohort 3b will receive HER3-DXd IV once every three weeks following an up-titration regimen (Cycle 1, Day 1: 57% of RDE or aRDE; Cycle 2, Day 1: 86% of RDE or, if applicable aRDE; Cycle 3 and subsequent cycles, Day 1: 114% of RDE or aRDE).
  Interventions: Drug: HER3-DXd (CTM-1 Lyo-DP)
- Dose Expansion: Cohort 4, EGFR mutant (Experimental): Participants with NSCLC (including any histology other than small-cell or combined small-cell and non-small cell) with an EGFR-activating mutation will receive HER3-DXd IV at 5.6 mg/kg every 3 weeks.
  Interventions: Drug: HER3-DXd (CTM-3 Lyo-DP)
- Dose Expansion: Cohort 5, KRAS-G12C mutant NSCLC (Experimental): Participants with locally advanced or metastatic NSCLC whose tumors harbor a KRAS-G12C mutation and that have progressed on the most recent line of therapy will receive HER3-DXd IV at 5.6 mg/kg every 3 weeks.
  Interventions: Drug: HER3-DXd (CTM-3 Lyo-DP)

INTERVENTIONS:
Drug: HER3-DXd (FL-DP) — HER3-DXd (frozen liquid drug product) consists of an antibody component (patritumab, U3-1287) covalently conjugated to a drug-linker (MAAA-1162a) containing a drug component (MAAA-1181a).
  Other Names: U3-1402
  Arms: Dose Escalation: Cohort 1, 3.2 mg/kg; Dose Escalation: Cohort 2, 4.8 mg/kg; Dose Escalation: Cohort 3, 5.6 mg/kg; Dose Escalation: Cohort 4, 6.4 mg/kg
Drug: HER3-DXd (CTM-1 Lyo-DP) — HER3-DXd (lyophilized drug product) consists of an antibody component (patritumab, U3-1287) covalently conjugated to a drug-linker (MAAA-1162a) containing a drug component (MAAA-1181a) that was manufactured by the clinical manufacturing sites.
  Other Names: U3-1402
  Arms: Dose Expansion: Cohort 1, EGFR mutant; Dose Expansion: Cohort 2, EGFR wild-type; Dose Expansion: Cohort 3a, EGFR mutant; Dose Expansion: Cohort 3b, EGFR mutant
Drug: HER3-DXd (CTM-3 Lyo-DP) — HER3-DXd (lyophilized drug product) consists of an antibody component (patritumab, U3-1287) covalently conjugated to a drug-linker (MAAA-1162a) containing a drug component (MAAA-1181a) that was manufactured by the commercial manufacturing sites.
  Other Names: U3-1402
  Arms: Dose Expansion: Cohort 4, EGFR mutant; Dose Expansion: Cohort 5, KRAS-G12C mutant NSCLC

SUMMARY:
This study was designed to evaluate safety and antitumor activity of HER3-DXd in two parts: Dose Escalation and Dose Expansion.

In Dose Escalation, HER3-DXd was evaluated in participants with metastatic or unresectable NSCLC with epidermal growth factor receptor (EGFR) activating mutation after disease progression during/after EGFR tyrosine kinase inhibitor (TKI) therapy.

In Dose Expansion, HER3-DXd will be evaluated in participants with metastatic or unresectable NSCLC with EGFR activating mutation or squamous or non-squamous NSCLC (ie, without EGFR-activating mutations) with disease progression during/after systemic treatment for locally advanced or metastatic disease.

In addition, HER3-DXd will be evaluated in participants with locally advanced or metastatic NSCLC whose tumors harbor a KRAS-G12C mutation after progression on the most recent line of therapy (Cohort 5).

DETAILED DESCRIPTION:
The primary objectives are:

* For Dose Escalation, to assess the safety and tolerability of HER3-DXd in the study population and to determine the recommended dose for expansion (RDE) of HER3-DXd in the study population
* For Dose Expansion, to investigate the antitumor activity of HER3-DXd
* For Cohort 5, investigate the antitumor activity of HER3-DXd in participants with locally advanced or metastatic NSCLC whose tumors harbor a KRAS-G12C mutation after the failure of targeted therapy

The number of treatment cycles is not fixed in this study. Participants will continue study treatment (for approximately 36 months) until they decide not to (withdraw consent), their disease gets worse [progressive disease (PD)], or side effects become unacceptable (unacceptable toxicity) or other stopping reasons have been met.

ELIGIBILITY:
Inclusion Criteria for both Dose Escalation and Dose Expansion:

1. Has locally advanced or metastatic NSCLC, not amenable to curative surgery or radiation
2. Has at least one measurable lesion per RECIST version 1.1
3. Has Eastern Cooperative Oncology Group performance status of 0 or 1 at Screening

Inclusion Criteria for Dose Escalation only:

1. Has histologically or cytologically documented adenocarcinoma NSCLC
2. Has acquired resistance to EGFR TKI according to the Jackman criteria (PMID: 19949011)

   1. Historical confirmation that the tumor harbors an epidermal growth factor receptor (EGFR) mutation known to be associated with EGFR tyrosine kinase inhibitor (TKI) sensitivity (including G719X, exon 19 deletion, L858R, L861Q)
   2. Has experienced clinical benefit from an EGFR TKI, followed by systemic progression of disease [Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1] or World Health Organization (WHO)] while on continuous treatment with an EGFR TKI
3. Is currently receiving and able to discontinue erlotinib, gefinitib, afatinib, or osimertinib
4. Has been receiving erlotinib, gefitinib, afatinib, or osimertinib for at least 6 weeks with well-controlled related toxicities less than Grade 3 in severity at the time of Screening
5. Has radiological documentation of disease progression while receiving continuous treatment with erlotinib, gefitinib, afatinib, or osimertinib
6. Is willing to provide archival tumor tissue from a biopsy performed within 6 months of progression during treatment with erlotinib, gefitinib, afatinib, or osimertinib OR has at least one lesion, not previously irradiated, amenable to core biopsy and is willing to undergo screening tumor biopsy
7. Demonstrates absence of EGFR T790M mutation if treated with erlotinib, gefitinib, or afatinib. No EGFR mutation testing is required if treated with osimertinib.

Inclusion Criteria for all cohorts of Dose Expansion only:

1. Has received systemic therapy for locally advanced or metastatic disease including at least 1 platinum-based chemotherapy regimen
2. Has documented radiological disease progression during/after most recent treatment regimen for locally-advanced or metastatic disease
3. For Cohorts 1, 2, 3a, and 3b: Is willing to provide archival tumor tissue from a biopsy performed within 6 months of consent and performed after progression during/after treatment with most recent cancer therapy regimen OR has at least 1 lesion, not previously irradiated, amenable to core biopsy and is willing to undergo tumor biopsy. Tumor tissue must be of sufficient quantity as defined in the laboratory manual and contain adequate tumor tissue content as confirmed by haematoxylin and eosin (H&S) staining at central laboratory.

   * For Cohort 4: Neither archival tumor tissue nor core tumor biopsy will be collected

Inclusion Criteria specific to Cohorts 1, 3a, 3b, and 4 of Dose Expansion:

1. Has histologically or cytologically documented:

   1. Cohort 1: Adenocarcinoma NSCLC
   2. Cohorts 3a, 3b, and 4: NSCLC (including any histology other than small-cell or combined small cell and non-small cell)
2. Has documentation of radiological disease progression following one or more lines of EGFR TKI treatment. Participants with EGFR T790M mutation following treatment with erlotinib, gefitinib afatinib, or dacomitinib must have received and have documentation of radiological disease progression following treatment with osimertinib unless unable or unwilling.
3. Has documentation of EGFR-activating mutation(s) detected from tumor tissue: G719X, exon deletion 19, L858R, or L861Q. Participants with other EGFR-activating mutations may be eligible following discussion with the Sponsor.

Inclusion Criteria specific to Cohort 2 of Dose Expansion:

1. Has histologically or cytologically documented squamous or non-squamous NSCLC (ie, without EGFR-activating mutations).
2. Has received prior treatment with anti-PD-1 or anti-PD-L1 antibody-based regimen in the locally advanced or metastatic setting unless unable or unwilling. Participants with NSCLC known to harbor a genomic alteration(s) other than EGFR mutation(s) (eg, ALK or ROS1 fusion) for which treatment is available must have also received prior treatment with at least 1 genotype-directed therapy.

Inclusion Criteria for Cohort 5:

1. Sign and date the main study ICF, prior to the start of any study-specific qualification procedures. A separate tissue screening consent will be obtained from all participants.
2. Male or female subjects aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old)
3. Has locally advanced or metastatic NSCLC not amenable to curative surgery or radiation.
4. Has histologically or cytologically documented squamous or nonsquamous NSCLC
5. Has documentation of KRAS-G12C mutation(s) detected from tumor tissue or liquid biopsy.
6. Has received at least two prior systemic therapies for locally advanced or metastatic disease, including 1 selective KRAS-G12C-targeted therapy (e.g., including as part of a clinical trial) (eg, the combination therapy of KRAS G12C-targeted therapy and immuno-oncology therapy can be considered as 2 prior systemic therapies).
7. Has documentation of radiological disease progression according to RECIST v1.1 while either on or following the most recent treatment regimen for locally advanced or metastatic disease.
8. Has ≥1 measurable lesion on computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST v1.1 by Investigator assessment that has not been previously irradiated.
9. Provides a pretreatment tumor tissue sample of sufficient quantity, as defined in the Study Laboratory Manual.
10. ECOG PS 0 or 1 at the time of Screening.
11. Has adequate bone marrow reserve and organ function based on local laboratory data within 14 days prior to Cycle 1 Day 1 as specified in the protocol.
12. If the participant is a female of childbearing potential, she must have a negative serum pregnancy test at screening and must be willing to use a highly effective birth control upon enrollment, during the Treatment Period, and for 7 months following the last dose of study drug.
13. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the time of final study drug administration.
14. If male, the subject must be surgically sterile or willing to use highly effective birth control upon enrollment, during the treatment period, and for at least 4 months following the last dose of study drug.
15. Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and for at least 4 months after the final study drug administration.
16. Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.

Exclusion Criteria for Dose Escalation and Dose Expansion:

1. Has any evidence of small cell histology, or combined small cell and non-small cell histology, in original tumor biopsy or in Screening biopsy performed after progression
2. Treatment with any of the following:

   1. Any cytotoxic chemotherapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than EGFR TKI in Cohorts 1, 3a, 3b, and 4 only), within 14 days of the first dose of study treatment
   2. Immune checkpoint inhibitor therapy within 21 days of the first dose of study treatment
   3. Prior treatment with an anti-HER3 antibody (dose escalation only)
   4. Prior treatment with a topoisomerase I inhibitor (dose escalation only)
   5. Prior treatment with an antibody-drug conjugate (ADC) that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, DS-8201a) (dose escalation only)
   6. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug treatment
   7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug treatment, or palliative radiation therapy within 2 weeks of the first dose of study drug treatment, or stereotactic radiotherapy within 1 week prior to the first dose of U3-1402
3. Has history of other active malignancy within 3 years prior to enrollment, except:

   1. Adequately treated non-melanoma skin cancer OR
   2. Superficial bladder tumors (Ta, Tis, T1) OR
   3. Curatively treated in situ disease
4. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study. Participants with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (1 week for stereotactic radiotherapy)
5. Has history of myocardial infarction within the past 6 months
6. Has symptomatic congestive heart failure[New York Heart Association (NYHA) Classes II-IV], unstable angina within the past 6 months, or cardiac arrhythmia requiring antiarrhythmic treatment
7. Has left ventricular ejection fraction (LVEF) < 50% by either echocardiogram (ECHO) or multigated acquisition scan (MUGA)
8. Has any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiogram (ECG), eg, complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval > 250 milliseconds (ms)
9. Has a mean corrected QT interval using Fridericia's Correction Formula (QTcF) prolongation to > 470 ms for females and > 450 ms for males in three successive Screening measurements
10. Unable or unwilling to discontinue concomitant drugs that are known to prolong the QT interval
11. Has any factors that increase the risk of corrected QT (QTc) interval prolongation or risk of arrhythmic events, such as congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
12. Has any history of interstitial lung disease (ILD) (including pulmonary fibrosis or severe radiation pneumonitis), has current ILD/pneumonitis, or is suspected to have such disease by imaging during screening
13. Has clinically significant corneal disease

Additional Exclusion Criteria for Dose Expansion Cohort 2:

1. Has documentation of one or more of the following EGFR-activating mutations: G719X, exon 19 deletion, L858R, or L861Q

Additional Exclusion Criteria for Dose Expansion Cohort 4:

1. Evidence of any leptomeningeal disease
2. Clinically severe respiratory compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

   1. Any underlying pulmonary disorder
   2. Any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement OR prior complete pneumonectomy
3. Is receiving chronic systemic corticosteroids dosed at >10 mg/day prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to enrollment
4. Resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
5. Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that could affect the safety of the subject; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results.

Exclusion Criteria for Cohort 5:

1. Has any evidence of small-cell histology or combined small cell and non-small-cell histology in the original tumor tissue or in Screening biopsy performed after progression.
2. Has received a targeted therapy for an actionable genomic alteration other than KRAS-G12C.
3. Has a history of interstitial lung disease (ILD)/pneumonitis) that required corticosteroid, has current ILD/pneumonitis, or wjhere suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
4. Has clinically severe respiratory compromise (based on the Investigator's assessment) resulting from intercurrent pulmonary illnesses.
5. Is receiving chronic systemic corticosteroids dosed at >10 mg/day prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1.
6. Has any history of or evidence of current leptomeningeal disease.
7. Has clinically significant corneal disease.
8. Evidence of spinal cord compression or brain metastases, defined as being clinically active and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
9. Inadequate washout period prior to Cycle 1 Day 1 as specified in the protocol.
10. Prior treatment with an anti-HER3 antibody and/or antibody drug conjugate (ADC) that consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, trastuzumab deruxtecan).
11. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute- Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0), Grade ≤1 or baseline.
12. Has known hypersensitivity to either the drug substance or inactive ingredients in the drug product.
13. Has history of other active malignancy within 3 years prior to Cycle 1 Day 1, with exceptions as specified in the protocol.
14. Uncontrolled or significant cardiovascular disorder prior to Cycle 1 Day 1,
15. Active Hepatitis B and/or Hepatitis C infection, such as that with serologic evidence of active viral infection within 28 days of enrollment.
16. Participants with past or resolved Hepatitis B virus (HBV) infection are eligible if meeting certain criteria as specified in the protocol.
17. Participants with a history of Hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks.
18. Has any evidence of severe or uncontrolled diseases, psychiatric illness/social situations, geographical factors, substance abuse, or other factors that, in the Investigator's opinion, make it high risk for the subject to participate in the study or that would jeopardize compliance with the protocol. Screening for chronic conditions is not required for eligibility.
19. Is a female participant who is pregnant or breastfeeding or intends to become pregnant during the study.
20. Has a known HIV infection that is not well controlled.
21. Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the participant; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) during dose escalation | 21 days of Cycle 1
Summary of adverse events during dose escalation | By the global end of trial date, approximately within 36 months
Overall response rate (ORR) assessed by Blinded Independent Central Review (BICR) Committee during dose expansion (Dose Expansion Cohorts 1, 2, 3a, 3b, and Cohort 5) | Approximately within 36 months
  ORR will be evaluated using RECIST v1.1.
Maximum serum concentration (Cmax) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose expansion (Cohort 4) | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Area under the serum concentration-time curve from time 0 extrapolated to infinity (AUCinf) and up to last quantifiable time (AUC[last]) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose expansion (Cohort 4) | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose escalation | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Time of maximum concentration (Tmax) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose escalation | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Area under the serum concentration-time curve from time 0 to 21 days (AUC[0-21]) and up to last quantifiable time (AUC[last]) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose escalation | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Overall response rate (ORR) during dose escalation | Approximately within 36 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) during dose escalation | Approximately within 36 months
Duration of response (DOR) during dose escalation | Approximately within 36 months
Time to response (TTR) during dose escalation | Approximately within 36 months
Progression free survival (PFS) during dose escalation | Approximately within 36 months
Overall Survival (OS) during dose escalation | Approximately within 36 months
Summary of adverse events during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | By the global end of trial date, approximately within 60 months
Maximum serum concentration (Cmax) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose expansion (Dose Expansion Cohorts 1-3 and Cohort 5) | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Time of maximum concentration (Tmax) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Area under the serum concentration-time curve from time 0 to 21 days (AUC[0-21]) and up to last quantifiable time (AUC[last]) of HER3-DXd, total anti-HER3 antibody, and MAAA-1181a during dose expansion (Dose Expansion Cohorts 1-3 and Cohort 5) | During the first 5 cycles (each cycle is 21 days), including an intensive sampling schedule: pre-dose, end of infusion (EOI), 2 hour (hr), 4 hr, 8 hr post infusion, Day 8, and Day 15.
Overall response rate (ORR) by Investigator during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
Duration of response (DOR) during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
Time to response (TTR) during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
Progression free survival (PFS) during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
Overall survival (OS) during dose expansion (Dose Expansion Cohorts 1-4 and Cohort 5) | Approximately within 60 months
Percentage of participants who are anti-drug antibody (ADA)-positive (baseline and post-baseline) and Percentage of participants who have treatment-emergent ADA during dose expansion (Cohort 4) | Approximately within 60 months
Mean Change from Baseline in the NSCLC-SAQ Total Score (Cohort 5) | Approximately within 60 months
  The NSCLC-SAQ will assess symptom severity over the previous 7 days. Participants will respond using a 5-point verbal rating scale ranging from 0 "No (symptom) at all" to 4 "Very severe (symptom)" or from 0 "Never" to 4 "Always". NSCLC-SAQ total score is the sum of 5 domains (cough, pain, dyspnea, fatigue, and poor appetite) and ranges between 0 and 20. Higher scores indicate more severe symptomatology. Mean change from baseline in NSCLC-SAQ total score will be reported.
Proportions of Deteriorated, Stable, or Improved Symptoms from NSCLC-SAQ (Cohort 5) | Approximately within 60 months
Proportions of Deteriorated, Stable, or Improved Symptoms from PRO-CTCAE (Cohort 5) | Approximately within 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Lead, Study Director — Daiichi Sankyo
Locations (37):
- United States (16):
  - City of Hope, Duarte, California
  - University of California San Diego, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - NYU Langone Health - NYU Medical Oncology Associates, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center (GCC) - Canton Facility, Canton, Ohio
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center (University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute/Tennesse Oncology, Nashville, Tennessee
  - Oncology Consultants P.A., Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Japan (5):
  - National Cancer Center Hospital East (NCCHE) - Kashiwa Campus, Kashiwa-Shi
  - Kurume University - Kurume University Hospital - Respiratory Diseases Center, Kurume-Shi
  - Kindai University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research (JFCR), Tokyo
- Netherlands Cancer Institute, Amsterdam, Netherlands
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - NEXT Oncology - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon (HGUGM), Madrid
  - Clinica Universidad Navarra(Madrid), Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Clínica Universidad de Navarra (Pamplona), Pamplona
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Jackman D, Pao W, Riely GJ, Engelman JA, Kris MG, Janne PA, Lynch T, Johnson BE, Miller VA. Clinical definition of acquired resistance to epidermal growth factor receptor tyrosine kinase inhibitors in non-small-cell lung cancer. J Clin Oncol. 2010 Jan 10;28(2):357-60. doi: 10.1200/JCO.2009.24.7049. Epub 2009 Nov 30. PMID 19949011
- [Derived] Steuer CE, Hayashi H, Su WC, Nishio M, Johnson ML, Kim DW, Massarelli E, Felip E, Gold KA, Murakami H, Baik CS, Kim SW, Smit EF, Fujimura M, Fan PD, Truchon K, Su X, Sternberg DW, Janne PA. Patritumab Deruxtecan (HER3-DXd; MK-1022) in Non-Small Cell Lung Cancer After Platinum-Based Chemotherapy and Immunotherapy. J Clin Oncol. 2025 Sep;43(25):2816-2826. doi: 10.1200/JCO-24-02744. Epub 2025 Jun 24. PMID 40554742